CLINICAL TRIAL: NCT04990336
Title: Comparison of Clinical Efficacy of Dachaihu Decoction Compound and Rhubarb Single Medicine in the Treatment of Acute Pancreatitis
Brief Title: Dachaihu Decoction Compound and Rhubarb Single Medicine in the Treatment of Acute Pancreatitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZDWY.XHNK.003
Record Dates: First submitted 2021-07-27; First posted 2021-08-04 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2021-07

CONDITIONS: Acute Pancreatitis
Keywords: Acute Pancreatitis; Dachaihu Decoction Compound; Rhubarb Single Medicine
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DDC(Dachaihu decoction compound) Group (Experimental): Treated with Dachaihu decoction compound and regular therapies
  Interventions: Combination Product: Dachaihu decoction compound; Combination Product: Regular therapies
- RSM(rhubarb single medicine) Group (Active Comparator): Treated with rhubarb single medicine and regular therapies
  Interventions: Drug: Rhubarb single medicine; Combination Product: Regular therapies
- N Group (Other): Treated with regular therapies and without traditional Chinese medicine
  Interventions: Combination Product: Regular therapies

INTERVENTIONS:
Combination Product: Dachaihu decoction compound — Dachaihu decoction compound includes Bupleurum, Rhubarb, Citrus aurantium, Scutellaria, Pinellia, White Peony, Jujube, Ginger.
  Arms: DDC(Dachaihu decoction compound) Group
Drug: Rhubarb single medicine — Rhubarb single medicine
  Arms: RSM(rhubarb single medicine) Group
Combination Product: Regular therapies — Regular therapies, such as fluid therapy, for acute pancreatitis

SUMMARY:
A large number of clinical studies have shown that oral administration, external application or enema of Chinese medicine can promote the recovery of gastrointestinal function and the absorption of pancreatic inflammation. The aims of the study is to explore the application of Dachaihu Decoction Compound (DDC)and Rhubarb Single Medicine (RSM) in the Treatment of Acute Pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years old
* Meet the diagnostic criteria of western medicine for acute pancreatitis, within 48 hours of onset
* Consent of the subjects, who sign the informed consent form

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Acute abdomen such as organic intestinal obstruction, gastrointestinal perforation, purulent cholangitis, etc.
* Patients with a history of severe heart, liver, kidney and other important organ diseases
* Patients with mental illness and malignant tumors
* People who have allergies, or are allergic to a certain drug ingredient

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Significant and effective rate | 7 days
  Significant and effective rate after 7 days of treatment